CLINICAL TRIAL: NCT02986412
Title: Evaluation of the Impact of a Topical Lotion, CG428, on Permanent Chemotherapy Induced Hair and Scalp Disorders in Cancer Survivors: An Open-label 6 Months Extension of VOLUME Study.
Brief Title: A 6-month Post-interventional Follow-up Extension of VOLUME Study (VOLUME-2)
Acronym: VOLUME2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Legacy Healthcare Services (Other)
Responsible Party: Principal Investigator, Juhee Cho, Chair, Assistant Professor Department of Clinical Research Design & Evaluation, SAIHST, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VOLUME2
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Alopecia; Chemotherapy Effects
MeSH Terms: conditions — Alopecia | interventions — CG428

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CG428 (Experimental): Patients will self-administer the study product twice per day (morning, evening) for 6 months, for the efficacy assessment
  Interventions: Other: CG428

INTERVENTIONS:
Other: CG428 — The experimental group will receive CG428. For each application, the patient should shake the bottle before spraying 10-12 times directly to the dry scalp whole area, with the nozzle, and then gently massage the whole scalp with fingertips in order to spread the lotion evenly until it has completely penetrated the scalp. Hairs should not be washed or shampooed within 1 hour following study treatment administration. Each dose should be spaced out by minimum 4 hours.

SUMMARY:
We would suggest to conduct "VOLUME-2" study, as an extension of the ongoing "VOLUME" study with all subjects already included. After completion of VOLUME study, the study will be directly extend with an "open-label design". All participants, who agreed to pursue, with either "Placebo" or "CG428", will receive CG428 treatment for an additional six-month period. VOLUME-2 study would be ideal and timely by enabling no interruption of product use.

The Primary Objective is to observe for a longer period the efficacy of CG428 (12 months : 6months Volume + 6 months Volume-2) in order to better discriminate later or non-responder populations.

Secondary Objectives are :

* Evaluate how far CG428 can improve hair-pattern (reach a plateau or constant progression)
* Evaluate motivation and adherence of subjects
* Long term safety

DETAILED DESCRIPTION:
The research team at Cancer Education Center at Samsung Comprehensive Cancer Center has studied CIA and its impact on distress and psychosocial well-being since 2008. We found that more than half of the breast cancer patients experienced higher distress due to CIA, during cancer treatment, and this distress was strongly associated with negative body image, overall health status, and psychosocial well-being. In a recent prospective cohort study, we assessed skin and hair change patterns before, during and 6 months after chemotherapy in 61 volunteers.

We found that the majority of the patients still experienced CIA at 6 months after completion of chemotherapy. Actually, hair diameter at 6th month after chemotherapy had not recovered to baseline level. Permanent chemotherapy-induced alopecia, defined as absent or incomplete hair regrowth at ≥6 months post-chemotherapy, was reported from 53 to 74%. Like CIA, permanent CIA also lacks recognition and has been underserved regardless of patients' needs. The first botanical blend Legacy Healthcare developed and patented is Cellium. Cellium is composed of 4 botanicals (Allium cepa L., Citrus limon L., Theobroma cacao L., Paullinia cupana).

The first product derived from Cellium is a topical lotion for male and female alopecia, CG210. Based on the safety and efficacy data, the EMA (European Medicines Agency) has considered CG210 eligible for a European centralized herbal medicine registration. CG428 is the second product derived from Cellium. CG428 contains the exact same ingredients as CG210, in a different dosage. Legacy Healthcare have conducted a pilot studies with CG428 in Japan. The trial included female cancer survivors experiencing permanent/persistent CIA for more than 12.

Based on the results, several cancer treatment centers in Japan have started to recommend the product on a compassionate basis.We therefore hypothesize that the investigated topical lotion may mitigate the impact of protracted or permanent CIA in cancer survivors by restoring a normalized apoptotic process of hair follicular cells and reducing the acute, as well as chronic inflammation in the scalp, two issues that may remain unsettled following anticancer treatment. While considering the subjects included in the "VOLUME" study, it appears that a majority of cancer survivors did not recover a full hair pattern even 3 years after cancer treatment. This is per se an interesting data, and a new and significant knowledge revealing that persistent chemotherapy induced apopecia (CIA) is more common than anticipated.

While considering the subjects included in the "VOLUME" study, it appears that a majority of cancer survivors did not recover a full hair pattern even 3 years after cancer treatment. This is per se an interesting data, and a new and significant knowledge revealing that persistent chemotherapy induced apopecia (CIA) is more common than anticipated.

The "VOLUME" study could have in fact two major repercussions: in addition to give information on CG428 efficacy, it will help to better define persistent CIA and improve thereby our scientific knowledge of this condition. Considering the high prevalence and poor literature on persistent CIA, it appears important to study this condition further.

To this end, we would suggest to conduct "VOLUME-2" study, as an extension of the ongoing "VOLUME" study with all subjects already included.

This study aims to evaluation of Longer observation (12 months : 6months Volume + 6 months Volume-2) permitting to better discriminate later or non-responder populations.

This is a open-label, single center, observation study in breast cancer survivors of VOLUME participants.

Hair condition and parameters of 31 breast cancer survivors who were previously included in VOLUME study (a randomized controlled trial to evaluate effect of CG428 which is topical hair lotion for chemotherapy induced alopecia completed in December, 2016) will be assessed.

The participation du extension Volume-2 study will be proposed to patients during the last visit of Volume study (Month 6)

The "VOLUME" study could have in fact two major repercussions: in addition to give information on CG428 efficacy, it will help to better define persistent CIA and improve thereby our scientific knowledge of this condition. Considering the high prevalence and poor literature on persistent CIA, it appears important to study this condition further.

To this end, we would suggest to conduct "VOLUME-2" study, as an extension of the ongoing "VOLUME" study with all subjects already included.

This study aims to evaluation of Longer observation (12 months : 6months Volume + 6 months Volume-2) permitting to better discriminate later or non-responder populations.

ELIGIBILITY:
Inclusion Criteria:

* hair parameters obtained before the start of chemotherapy
* Patients who participated in VOLUME
* Able to keep their hair style
* Able to use the study treatment in compliance with the protocol.
* Physical (ECOG≤1) and psychological ability to participate

Exclusion Criteria:

* Concomitant use of other anti-hair-loss treatment or hair growth treatment.
* Patients with recent hair transplants or who plan to have transplants.
* Known allergy or hypersensitivity to some components of CG428 (including allium cepa (onion), citrus, caffeine, theobromine)
* Pre-existing alopecia or significant scalp disease, which may alter study treatment administration or absorption.

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Hair thickness | 6 months after intervention
  Objectively quantified hair thickness will measure using Folliscope 4.0, LeadM

SECONDARY OUTCOMES:
Chemotherapy-induced alopecia distress Stress Using Chemotherapy induced | All time (baseline, 3month and 6 months after intervention)
  Respondents will be instructed to indicate on a 4-point Likert scale on each
Global photographs | All time (baseline, 3month and 6 months after intervention)
  Pictures to be focused on head/hair, which means shorter distance between the equipment and the subject using Canon EOS 70D
Overall hair and scalp condition | All time (baseline, 3month and 6 months after intervention)
  Patient self-assessment: We will use self-reported questionnaire using visual analogue scale (VAS) ranging from 0 to 10.
Nail condition | All time (baseline, 3month and 6 months after intervention)
  Patient self-assessment: We will use self-reported questionnaire using visual analogue scale (VAS) ranging from 0 to 10.
Quality of life at the time | All time (baseline, 3month and 6 months after intervention)
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 and breast specific module
Satisfaction with products | All time (baseline, 3month and 6 months after intervention)
  We will use self-reported questionnaire for satisfaction with the products as well as suggestions for improvement after completion of study with patients who received the CG428.
Willing to Pay | 6 months after intervention
  We will ask how much to willing to pay for CG428
Hair condition | All time (baseline, 3month and 6 months after intervention)
  Outcomes will be collected using objective methods and patient reported outcomes:
  Objectively quantified: Hair thickness and density: We will measure hair thickness and density using Folliscope 4.0, LeadM We will take a picture on the parietal (To around 2 cm) and then analysis using Folliscope program.
  Global photographs: Pictures to be focused on head/hair, which means shorter distance between the equipment and the subject

OTHER OUTCOMES:
Group in VOLUME | At baseline
  Information about what group they belonged to in previous studies

CONTACTS AND LOCATIONS:
Overall Officials: Juhee Cho, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Danbee Kang, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: EValuation of the Impact of a TOpical Lotion on Permanent Chemotherapy Induced Hair Disorders in Cancer Survivors (VOLUME) — https://clinicaltrials.gov/ct2/show/NCT02605629?term=juhee+cho&rank=1